CLINICAL TRIAL: NCT06793696
Title: Adaptive Decision Support for Addiction Treatment (ADAPT) Factorial Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2000038624-A; 5R33DA059884-02 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder; Clinical Decision Support
Keywords: Opioid use disorder; clinical decision support
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Eligible patients are randomized to a study arm during Emergency Department encounters at study sites. There is no open enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- EMBED CDS (Active Comparator): Provider receives EMBED CDS
  Interventions: Other: EMBED
- EMBED CDS and nurse prompt (Experimental): EMBED CDS and nurse receives prompt to complete COWS
  Interventions: Other: Nurse prompt; Other: EMBED
- EMBED CDS and provider prompt (Experimental): EMBED CDS and provider prompt for EMBED CDS
  Interventions: Other: Provider prompt; Other: EMBED
- EMBED CDS and patient facing materials (Experimental): EMBED CDS and patient materials at patient discharge from ED
  Interventions: Other: Patient facing materials; Other: EMBED
- EMBED CDS and nurse prompt and provider prompt (Experimental): EMBED CDS and nurse prompt to complete COWS and provider prompt for CDS
  Interventions: Other: Nurse prompt; Other: Provider prompt; Other: EMBED
- EMBED CDS and nurse prompt and patient facing materials (Experimental): EMBED CDS and nurse prompt to complete COWS and patient materials at discharge from ED
  Interventions: Other: Nurse prompt; Other: Patient facing materials; Other: EMBED
- EMBED CDS and provider prompt and patient facing materials (Experimental): EMBED CDS and provider prompt for EMBED and patient materials at discharge from ED
  Interventions: Other: Provider prompt; Other: Patient facing materials; Other: EMBED
- EMBED CDS and nurse prompt and provider prompt and patient facing materials (Experimental): EMBED CDS and nurse prompt to complete COWS and provider prompt to complete CDS and patient materials at discharge from ED
  Interventions: Other: Nurse prompt; Other: Provider prompt; Other: Patient facing materials; Other: EMBED

INTERVENTIONS:
Other: Nurse prompt — Nurse prompt to complete COWS
  Arms: EMBED CDS and nurse prompt; EMBED CDS and nurse prompt and patient facing materials; EMBED CDS and nurse prompt and provider prompt; EMBED CDS and nurse prompt and provider prompt and patient facing materials
Other: Provider prompt — Provider prompt to use EMBED CDS
  Arms: EMBED CDS and nurse prompt and provider prompt; EMBED CDS and nurse prompt and provider prompt and patient facing materials; EMBED CDS and provider prompt; EMBED CDS and provider prompt and patient facing materials
Other: Patient facing materials — Patient materials provided at discharge from ED
  Arms: EMBED CDS and nurse prompt and patient facing materials; EMBED CDS and nurse prompt and provider prompt and patient facing materials; EMBED CDS and patient facing materials; EMBED CDS and provider prompt and patient facing materials
Other: EMBED — Original EMBED CDS

SUMMARY:
This study is stage 1 of a larger study which refines and optimizes the EMBED* clinical decision support (CDS; see NCT03658642) to increase number of ED physicians following standard of care for the administration of buprenorphine to appropriate patients with opioid use disorder.

This study does not have open enrollment. Investigators will use a Multiphase Optimization STrategy (MOST) framework study with preparation, optimization, and confirmatory phases. In the current project, optimization phase, stage1 investigators will conduct a 2x2x2 factorial trial in which they expand EMBED to include sustainable implementation strategies: nurse prompt for withdrawal assessment, and targeted clinician prompt to use the CDS along with patient resources to promote equity and motivate readiness to start treatment.

Later study phases will include optimization phase, stage 2: rapid-cycle randomized testing, and evaluation phase: a randomized trial of the optimized package compared to the original EMBED and the evaluation phase in which investigators will compare the efficacy of the optimized, multicomponent CDS package to the original EMBED CDS on ED-initiation of buprenorphine rates in patients with OUD in a randomized trial.

*EMBED is a user centered, clinician facing clinical decision support system integrated into the electronic health record workflow to facilitate initiating buprenorphine in the emergency department by: diagnosing opioid use disorder with a checklist based on the diagnostic criteria of the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, fifth edition), assessing the severity of withdrawal with the Clinical Opioid Withdrawal Scale (COWS), motivating patients to accept treatment with a scripted brief negotiation interview, and automating the electronic health record workflow, including clinical and after visit documentation, order entry, prescribing, and referral for ongoing treatment in the community

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patient
* 18 years of age or older
* Moderate to severe opioid use disorder

Exclusion Criteria:

* Under 18 years of age
* Pregnant
* Currently receiving medication for opioid use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1129 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of encounters with Buprenorphine initiation in the ED | Upon discharge from the ED, 1 day
  Proportion of eligible encounters with buprenorphine administered in the Emergency Department (ED) and/or prescribed buprenorphine on discharge from the ED. Obtained from EHR data.
Proportion of alerted encounters with CDS engagement | Trial start to end up to 18 months
  Proportion of eligible encounters in the Emergency Department with an alert fired (silent or active) with CDS engagement. CDS engagement is defined as: OUD diagnosis entered via CDS, withdrawal assessment, readiness assessment, buprenorphine order/prescription placed, referral placed, or any flowsheet item completed.

SECONDARY OUTCOMES:
Proportion of encounters with Naloxone prescription upon ED discharge | Upon discharge from the ED, 1 day
  Proportion of eligible encounters with naloxone prescribed on discharge from the Emergency Department (ED). Obtained from EHR data.
Proportion of encounters with patient referral to ongoing MOUD treatment | Upon discharge from the ED, 1 day
  Proportion of eligible encounters with referral for ongoing MOUD treatment received on discharge from the Emergency Department (ED). Obtained from EHR data.
Proportion of encounters with patient receipt of appropriate opioid related discharge instructions | Upon discharge from the ED, 1 day
  Proportion of encounters with appropriate opioid related discharge instructions. Obtained from EHR data.
Proportion of attending physicians initiating BUP in the ED for at least one eligible patient | Trial start to end up to 18 months
  Proportion of attending physicians administered or prescribed Buprenorphine in the Emergency Department (ED) for at least one encounter. Obtained from EHR data.
Proportion of attending physician prescribing naloxone upon ED discharge | Trial start to end up to18 months
  Proportion of attending physicians prescribing naloxone in the Emergency Department (ED) for at least one encounter. Obtained from EHR data.
Proportion of attending physician referral to ongoing MOUD treatment | Trial start to end up to 18 months
  Proportion of attending physicians referring a patient to ongoing MOUD treatment on discharge from the Emergency Department (ED) for at least one encounter. Obtained from EHR data.
Proportion of attending physicians giving appropriate opioid related discharge instructions | Trial start to end up to 18 months
  Proportion of attending physicians giving appropriate opioid related discharge instructions for at least one encounter. Obtained from EHR data.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Melnick, MD, MHS, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale New Haven Shoreline Medical Center, Guilford, Connecticut
  - Yale New Haven Hospital- St. Raphael, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to EHR use measurements in various levels of aggregation. e.g., time spent on the CDS or threshold outcomes such as dismissal of the CDS without action under a specific amount of time or the time spent on CDS that exceeds what was expected based on the patient's clinical opioid withdrawal (COWS) score, time in the ED, or level of acuity, patient acuity, chief complaints or diagnoses, clinician, interruptions (such as orders started but not finished), task switching, seasonality, and variation in shift timing (such as nights and weekends). Data shared will include variables relating to patient demographics, medical history, prescription information, clinician facing clinical decision support (CDS) firing and clinician action information, and clinician prescribing decisions and historical prescribing
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified data will be shared with NAHDAP as soon as possible upon completion of quality control procedures, analysis, and at the time of associated publication or end of performance period. Data will be released by NAHDAP at the time of receipt and will be available indefinitely
Access Criteria: De-identified data sets used for analysis will be submitted to NAHDAP through the NIH HEAL Initiative and will be available for public use according to NAHDAP data sharing policies and restrictions set by our DUA with NAHDAP and our IRB. All data submissions to NAHDAP undergo confidentiality review to protect respondents' data from being re-identified.
  Portions of the ADAPT intervention will be built for national distribution on the Epic EHR platform. Distribution of code that is proprietary to Epic may limit distribution of certain portions of software or code. In this situation, investigators will provide dashboards and visualizations of workflow diagrams as appropriate to disclose interface and workflow concepts to the broader scientific community These portions of the data will also be subject to restricted use access outside of organizations using Epic.